CLINICAL TRIAL: NCT01766544
Title: Asthma and COPD Guideline Implementation: Lessons Learned on Recruitment of Primary Care Physicians to a Knowledge Translation Study
Brief Title: Asthma & COPD Guideline Implementation
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment of physicians to participate to the study.
Sponsor: Laval University (Other)
Collaborators: GlaxoSmithKline (Industry); Canadian Lung Association (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: GIPC
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Last update posted 2013-01-11 (Estimated); Status verified 2013-01

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: asthma; COPD; guidelines; knowledge transfer; medical education; care gaps
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard practice group (SPG) (Active Comparator): Send a copy of the latest Canadian asthma and COPD guidelines to all PCPs.
  Interventions: Other: Standard Practice Group (SPG)
- Targeted Intervention Strategy (TISG) (Active Comparator): interactive educational intervention, expert mentorship, practice-based tools. Consisting of 3 interactive sessions, 2 of which would be live meetings of 3h each and the third a one-hour teleconference.
  Interventions: Other: TISG

INTERVENTIONS:
Other: Standard Practice Group (SPG) — The investigators planned to send a copy of the latest Canadian asthma and COPD guidelines to all PCPs in the Standard Practice (SP) Group at the start of the study period, by mail. No other intervention would be offered during the study, but upon study completion, all control participants would be offered the educational intervention received by the Targeted Intervention Strategy (TIS) Group.
  Arms: Standard practice group (SPG)
Other: TISG — interactive educational interventions, expert mentorship and practice-based tools. 3 interactive sessions, 2 of which would be live meetings of 3h each, and the third hour teleconference.
  Arms: Targeted Intervention Strategy (TISG)

SUMMARY:
This is a report of a protocol developed to improve asthma and COPD care in a primary care setting. The study was approved by an Ethics Committee and support by the Canadian Thoracic Society through an unrestrictive grant from GlaxoSmithKline. However, the study could not be done and the investigators report why, discussing the difficulties to perform such study. This information should be very useful to investigators planning this sort of study.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are the two most common chronic pulmonary ailments in Canada, affecting about 2.5 million and 750 thousand individuals, respectively. In the last two decades, the Canadian Thoracic Society (CTS) has successfully developed and disseminated evidence-based asthma and COPD clinical practice guidelines. However, evidence suggests that guideline implementation in these diseases remains inadequate.

Successful guideline implementation requires tailoring of selected strategies to settings and population-specific barriers, based on established theories and principles. In 2004, the CTS and its collaborators organized a symposium in Quebec City, to discuss existing barriers to respiratory guideline implementation and possible knowledge translation (KT) strategies. This was followed in the fall of 2007 by an expert-led workshop on guideline implementation strategies.

Herein, the investigators report the planned methods and outcome of a project which resulted from these meetings. This study sought to explore the effectiveness of a multi-faceted KT strategy in improving concordance with COPD and asthma guidelines among primary care physicians (PCPs) in Canada, but was aborted due to inadequate PCP recruitment. The investigators discuss the difficulties encountered in recruiting PCPs, factors which may have influenced recruitment, and alternative strategies. The goal of the investigators is to provide practical lessons to inform the design of future KT initiatives with similar interventions and/or a similar target audience.

ELIGIBILITY:
Inclusion Criteria:

Primary care physicians were eligible if they: 1) managed at least 15 patients with asthma and 15 patients with COPD per month in an office setting; and 2) agreed to designate an appropriately trained person at his/her site to identify eligible study patients, collect consent, and provide a questionnaire to patients.

Patients were eligible if they: 1) spoke French or English; and 2) had a diagnosis of asthma or COPD (as per their participating PCP). Furthermore, patients with asthma had to be between 18 and 45 years of age, and patients with COPD had to be between 40 and 75 years of age and have a smoking history of >10 pack-years.

Exclusion Criteria:

Physicians were excluded if they: 1) had presented at a continuing medical education (CME) event on asthma or COPD in last year; 2) had completed any specialty training in respiratory diseases; or 3) practiced primarily at walk-in clinics, with children, or in emergency departments.

Patients were excluded if they: 1) had any condition which could interfere with study measurements (as per their participating PCP); 2) had any known respiratory disorders other than asthma or COPD; or 3) were currently participating in another clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Physician Assessment Questionnaire-Asthma | First visit
  The co-primary outcomes (for asthma and COPD) were defined as the change in patient-reported physician conformity to each of the following key guideline recommendations, measured through a questionnaire (Appendix 1):
  A) For asthma, assessment of asthma control, defined as ascertainment of at least 2 of the 5 asthma control questions recommended by the Canadian Asthma Guidelines. Stratified physician randomization would randomize 75% of PCPs to the TIS group and 25% to the SP group.

SECONDARY OUTCOMES:
The Physician Practice Assessment Questionnaire | First visit
  Secondary outcomes collected through the patient questionnaires included other guideline-recommended physician behaviours. For asthma, these included spirometry performance, asthma action plan provision and review, inhaler technique review, and maintenance anti-inflammatory medication prescription when indicated. For COPD, these included spirometry performance, inhaler technique review, exacerbation screening, long-acting bronchodilator prescription when indicated, and smoking cessation efforts in smokers. A separate questionnaire measured physician self-reported changes in knowledge and adherence to guideline-recommended behaviours (the "Physician Practice Assessment Questionnaire") (PPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Boulet, MD, FRCPC, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada